CLINICAL TRIAL: NCT01486576
Title: Effect of Hydroxyethyl Starch on Renal Handling of Sodium and Water, Vasoactive Hormones,Biomarkers and the Circulatory System in Patients Undergoing Hip Replacement Surgery
Brief Title: Hydroxyethyl Starch and Renal Function After Hip Replacement Surgery
Acronym: VOHO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASK-3-2011
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — HES 130-0.4; Hydroxyethyl Starch Derivatives; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voluven (Hydroxyethyl starch 130/0,4) (Active Comparator): Patients undergoing hip replacement surgery will receive either fluid therapy with active comparator (Voluven) or placebo (Sodium Chloride. Patients will receive minimum 7,5 ml/kg in the first hour of the surgery and 5 ml/kg in the subsequent hours.
  Interventions: Drug: Voluven (Hydroxyethyl starch 130/0,4)
- Sodium Chloride 9 mg/ml (Placebo Comparator): Patients undergoing hip replacement surgery will receive either fluid therapy with active comparator (Voluven) or placebo (Sodium Chloride. Patients will receive minimum 7,5 ml/kg in the first hour of the surgery and 5 ml/kg in the subsequent hours.
  Interventions: Drug: Sodium Chloride 9 mg/ml

INTERVENTIONS:
Drug: Voluven (Hydroxyethyl starch 130/0,4) — 7,5 ml/kg in the first hour and then 5 ml/kg
  Other Names: Voluven; Venofundin; Hydroxyethyl starch
  Arms: Voluven (Hydroxyethyl starch 130/0,4)
Drug: Sodium Chloride 9 mg/ml — 7,5 ml/kg in the first hour and then 5 ml/kg
  Other Names: Isotone saline solution
  Arms: Sodium Chloride 9 mg/ml

SUMMARY:
The purpose of this project is to investigate if hydroxyethyl starch (HES) is potential nephrotoxic and examine the effects on the circulation and kidneys during administration of HES during surgery.

DETAILED DESCRIPTION:
Hydroxyethyl starch (HES) is widely used in hospitals to maintain circulation in critically ill patients. In recent years studies have raised suspicion that HES is nephrotoxic. So far acute kidney injury has been diagnosed based on creatinine measurements, but new technology allows for earlier diagnosis using measurements of biomarkers in urine.

The purpose of this project is to investigate HES's potential toxicity and effects on the circulation and kidneys using measurements of biomarkers specific for toxicity and for the sodium/water balance in the urine and by measurements of vasoactive hormones in the blood after administration of HES 130/0.4

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Males and females
* Indication for Arthroplasty of hip

Exclusion Criteria:

* Blood donation within the last month
* Lack of wish to participate
* eGFR< 15ml/min
* pregnancy or breast feeding
* Need of NSAID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
u-NGAL | 2-4 hours
  The main objective is for the trial (only patients undergoing elective hip replacement surgery) to measure the effect of hydroxyethyl starch on u-NGAL, which is a biomarker of nephrotoxicity

SECONDARY OUTCOMES:
u-Kim1, u-LFABP | 2-4 hours
  Another objective of the trial (only patients undergoing elective hip replacement surgery) to measure the effect of hydroxyethyl starch on u-Kim1 and u-LFABP, which are biomarkers of nephrotoxicity
FENa, u-ENaCβ, CH2O, u-AQP2,u-NCC, u-NK2CC | 2-4 hours
  Secondarily to measure the effect of hydroxyethyl starch on the renal tubular transport of sodium and water during elective hip replacement surgery
PRC, p-Ang-II, p -Aldo, p-ANP,P-GDP, p-AVP, p-Endot | 2-4 hours
  Secondarily to measure the effect of hydroxyethyl starch on vasoactive hormones during elective hip replacement surgery
SBP, DBP, heartrate | 2-4 hours
  Secondarily to measure the effect of hydroxyethyl starch on central hemodynamics during elective hip replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie P. Kancir, MD PhD, Principal Investigator — Holstebo Regional Hospital
Locations (1):
- Medicinsk forskningsafsnit, Regionshospitalet Holstebro, Holstebro, Denmark